CLINICAL TRIAL: NCT07142148
Title: Validation of the Celiac Dietary Adherence Test in the Polish Paediatric Population
Brief Title: Validation of the CDAT in the Polish Paediatric Population
Acronym: CD-PL-CDAT
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Aleksandra Banaszkiewicz, MD, PhD, Prof., Medical University of Warsaw
Other Study IDs: CD-PL-CDAT
Record Dates: First submitted 2025-08-18; First posted 2025-08-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Coeliac Disease; Celiac Disease in Children
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CDAT - phase 1 — The English version of the Celiac Dietary Adherence Test (CDAT) will be translated into Polish using the "forward-backwards-forward" translation model, with the author's consent (already obtained by the applicants). The Polish translation will be performed by two native bilingual speakers of Polish and English. Both translations will be compared and standardised. The Polish version will then be translated into English by two native bilingual speakers of English who are unfamiliar with the original English version. The translation and original will be compared to clarify discrepancies and ensure conceptual equivalence between the versions. The agreed-upon translation will be culturally adapted, if necessary. The items will be reviewed by five experts, and an I-CVI of at least 0.78 will be considered satisfactory content validity.
Other: CDAT - phase 2 — In the next step, 10 coeliac disease (CD) patients aged 10 years and older and 10 caregivers/parents of CD patients under 10 years of age will be asked to rate the clarity of each statement on a Likert scale [1 = unclear to 5 = very clear]. Questions with a mean score <4.0 will be rephrased and re-evaluated.
  Internal consistency analysis using Cronbach's alpha and the mean inter-item correlation (AIC) will be used to assess reliability. Convergent validity will be assessed by comparing scale scores with serological marker levels. Confirmatory factor analysis (CFA) will be conducted, taking into account the SRMR fit index.

SUMMARY:
The English version of the Celiac Dietary Adherence Test (CDAT) will be translated into Polish using the "forward-backwards-forward" translation model, with the author's consent (already obtained by the applicants).

The Polish translation will be performed by two native bilingual speakers of Polish and English. Both translations will be compared and standardised. The Polish version will then be translated into English by two native bilingual speakers of English who are unfamiliar with the original English version. The translation and original will be compared to clarify discrepancies and ensure conceptual equivalence between the versions. The agreed-upon translation will be culturally adapted, if necessary. The items will be reviewed by five experts, and an I-CVI of at least 0.78 will be considered satisfactory content validity.

In the next step, 10 coeliac disease (CD) patients aged 10 years and older and 10 caregivers/parents of CD patients under 10 years of age will be asked to rate the clarity of each statement on a Likert scale [1 = unclear to 5 = very clear]. Questions with a mean score <4.0 will be rephrased and re-evaluated.

Internal consistency analysis using Cronbach's alpha and the mean inter-item correlation (AIC) will be used to assess reliability. Convergent validity will be assessed by comparing scale scores with serological marker levels. Confirmatory factor analysis (CFA) will be conducted, taking into account the SRMR fit index.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of coeliac disease (CD) according to the European Society of Pediatric Gastroenterology and Nutrition (ESPGHAN) criteria,
* age from 2 to 18 years of age,
* consent from legal guardians (and the child in case of patients ≥16 years of age) to participate in the study.

Exclusion Criteria:

* whose legal guardians did not consent to participate in the study,
* who did not consent to participate in the study (applies to patients ≥ 16 years of age).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Polish children with CD.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Validation of Celiac Dietary Adherence Test (CDAT) in the Polish paediatric population. | September 2025 - June 2027
  The Celiac Dietary Adherence Test (CDAT) questionnaire will be validated in the Polish paediatric population.